CLINICAL TRIAL: NCT06257771
Title: Pharmacokinetics and Responses to Alcohol After Bariatric Surgery
Brief Title: Alcohol After Bariatric Surgery 2
Acronym: ABS2
Status: Recruiting | Type: Observational
Sponsor: University of Illinois at Urbana-Champaign (Other)
Collaborators: Carle Foundation Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 24444 (old); IRB24-0173 (new)
Record Dates: First submitted 2024-02-05; First posted 2024-02-14 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Sleeve Gastrectomy
Keywords: Alcohol metabolism; Bariatric surgery; Hypoglycemia; Metabolic surgery
MeSH Terms: conditions — Hypoglycemia | interventions — Ethanol

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Women 1-5 years post-SG: * Alcohol orally administered (0.5 grams per kg of Fat-free mass) after overnight fast or after a standard meal
  * Alcohol administered IV using an alcohol clamp (target concentration of 0.6g/L after an overnight fast or one hour after consuming a standard mixed meal)
  Interventions: Drug: Alcohol (Ethanol)
- Men 1-5 years post-SG: * Alcohol orally administered (0.5 grams per kg of Fat-free mass) after overnight fast or after a standard meal
  * Alcohol administered IV using an alcohol clamp (target concentration of 0.6g/L after an overnight fast or one hour after consuming a standard mixed meal)
  Interventions: Drug: Alcohol (Ethanol)
- Women, non-operated control: * Alcohol orally administered (0.5 grams per kg of Fat-free mass) after overnight fast or after a standard meal
  * Alcohol administered IV using an alcohol clamp (target concentration of 0.6g/L after an overnight fast or one hour after consuming a standard mixed meal)
  Interventions: Drug: Alcohol (Ethanol)
- Men, non-operated control: * Alcohol orally administered (0.5 grams per kg of Fat-free mass) after overnight fast or after a standard meal
  * Alcohol administered IV using an alcohol clamp (target concentration of 0.6g/L after an overnight fast or one hour after consuming a standard mixed meal)
  Interventions: Drug: Alcohol (Ethanol)

INTERVENTIONS:
Drug: Alcohol (Ethanol) — Alcohol given orally (0.5 grams of alcohol per kg of fat-free mass) Alcohol given iv with a clamp ( 6% v/v alcohol prepared in 0.5% normal saline). The infusion rate will exponentially increase from the start of the infusion until the target BrAC of 0.6g/L (60mg%) is reached at 15 min, followed by an exponentially decreasing infusion rate, which will be tapered to a constant steady-state value to clamp the BrAC at the target value for a predetermined duration of 180 min.

SUMMARY:
The goal of this observational study is to learn how the body processes ingested alcohol and how alcohol affects mood and blood sugar in both men and women after undergoing sleeve gastrectomy. The main question[s]it aims to answer are:

* Are there differences in the way that ingested alcohol is handled in men versus women after sleeve gastrectomy?
* What is the consequence of drinking alcohol on an empty stomach versus after a meal on blood sugar control after undergoing sleeve gastrectomy?

Participants will participate in two types of alcohol tests (alcohol given orally or administered intravenously) after not eating anything overnight or after having a meal.

Researchers will compare men and women who underwent sleeve gastrectomy with men and women who had no surgery, are of similar age and body composition, and have similar alcohol intake patterns.

DETAILED DESCRIPTION:
The primary goal of the proposed study is to determine sex-related differences in the impact of Sleeve Gastrectomy (SG) on the pharmacokinetics (Aim 1), subjective effects (Aim 2), and glycemic effects (Aim 3) in the fasted versus prandial state when alcohol is ingested or given intravenously clamped (the gold standard to measure alcohol elimination rate and acute alcohol tolerance). We will use a cross-sectional study to compare participants who underwent SG surgery 1-5 years ago with matched non-operated controls (both sexes). This project will answer the questions of whether there are sex-related differences in the impact of SG on alcohol's pharmacokinetics and pharmacologic effects, whether drinking alcohol with a meal is effective post-SG, and clarify the site of alcohol first-pass metabolism in men. Findings from this study will contribute to evidence-based recommendations on the impact of SG on alcohol-related toxic effects and could help expand the knowledge base of sex-related differences in human alcohol pharmacokinetics.

ELIGIBILITY:
Inclusion Criteria:

* Surgery groups:

  * Male and female, 21-64 yrs. of age
  * Drink at least 1 standard drink per month but no more than 7 per week (women or > 14 for men)
  * Underwent SG surgery 1-5 years ago

Non-surgery control group

* Male and female who did not undergo bariatric surgery
* Age , BMI, race , and alcohol pattern of consumption equivalent to participants in the SG surgery groups

Exclusion Criteria:

* For all groups (surgery and non-surgery groups)

  * Smoking or having quit smoking less than 2 months ago
  * Pregnant or breastfeeding
  * Taking any medications that might affect alcohol metabolism
  * Anemia
  * Gastritis, colitis, Crohn's Disease, malabsorptive diseases, inflammatory diseases, liver disease, kidney disease, cancer less than five years ago, stroke, or severe organ dysfunction
  * Body weight >450 pounds (because of a limit on body composition machine)
  * Alcohol use disorder
  * Regular use of drugs with addiction potential or regular misuse of substances
  * Abnormality on EKG as determined by a study physician to present a safety risk

Ages: 21 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Carle Foundation Hospital and community sample
Sampling Method: Non-Probability Sample
Enrollment: 88 (Estimated)
Dates: Start 2024-07-31 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Blood alcohol concentrations (BAC) | From zero to up to 180 minutes post alcohol administration
  The concentration of alcohol measured in arterialized venous blood and estimated from breath )BrAC)
Subjective effects of alcohol | Before and after (10-180 min) they consume the alcoholic beverage or receive the IV infusion for the alcohol clamp.
  We will use valid psychometrically sound instruments to assess alcohol's subjective effects (e.g., stimulant and sedative effects of alcohol)
Plasma glucose concentrations | Before and after (10-180 min) they consume the alcoholic beverage.
  The concentration of glucose measured in plasma.

SECONDARY OUTCOMES:
Gut hormones and other peptides | Before and after (10-180 min) they consume the alcoholic beverage
  Gut hormones such as ghrelin, glucagon-like peptide and others

CONTACTS AND LOCATIONS:
Overall Officials: Marta Y Pepino de Gruev, PhD, Principal Investigator — University of Illinois at Urbana-Champaign
Locations (1):
- University of Illinois at Urbana Champaign, Urbana, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be findable for the research community through NIAAADA. The research community will have access to data at the time of publication or when the award ends, whichever is sooner. NIAAADA will make decisions about how long to preserve the data.
Supporting Information: ICF
Time Frame: The research community will have access to data at the time of publication or when the award ends, whichever is sooner. NIAAADA will make decisions about how long to preserve the data.
Access Criteria: To request access of the data, researchers will use the standard processes at NIMH Data Archive (NDA) , and the NDA Data Access Committee will decide which requests to grant. The standard NDA data access process allows access for one year and is renewable